CLINICAL TRIAL: NCT03036436
Title: Investigating the Feasibility and Acceptability of a Technology Delivered Physical Activity (PA) Intervention in Cancer: The IMPETUS Cancer Trial. (IMproving Physical Activity and Exercise With Technology Use in Cancer Survivors)
Brief Title: The IMPETUS Cancer Trial. A Technology Delivered Physical Activity Intervention in Cancer
Acronym: IMPETUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Ciaran Haberlin, PhD Candidate, Chartered Physiotherapist, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IMPETUS-01
Record Dates: First submitted 2016-12-19; First posted 2017-01-30 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Cancer, Breast; Cancer, Colorectal; Malignancy
Keywords: Cancer; EHealth; Cancer Survivor; Rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participants in this group will receive the intervention. They will receive a Fitbit activity tracker, and will also receive support and goal setting with a view to improving their daily physical activity.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — A physical activity intervention, delivered remotely using a combination of the Fitbit application and support from a chartered physiotherapist.

SUMMARY:
Participants will take part in a 12 week intervention, with at least one follow up at 24 +/- 2 weeks. Each participant will be provided with support, motivation and professional guidance about improving physical activity (PA) levels and will be given a commercially available PA tracker. The PA tracker will also include a smartphone or web-based application, where participants can upload their exercise performed each day, and keep up to date with their goals using their smartphone or by logging on to their computer. The aim of the study is to find out how useful and effective technology with support from a healthcare professional is in helping cancer survivors to become more physically active.

This study will measure objective PA levels of the participants at the start of the study and at the end. The acceptability of using this intervention to promote PA in cancer survivors will also be investigated.

DETAILED DESCRIPTION:
The overall aim is to determine the feasibility of a specific PA intervention, combining technology and professional input, in the cancer survivor population.

Study Design: A single arm feasibility trial of a PA intervention using technology and behavioural change theories as tools to achieve increased PA. Participants in the study will receive 12 weeks of the intervention. Outcomes will be measured at baseline, 12 weeks and 24 weeks (+/- 2 weeks) post baseline.

Patient recruitment: Participants will be recruited from those attending the St. James' Hospital oncology and haematology services. Study personnel will provide further information to these patients and assess them for eligibility. Informed consent will be gained from each participant.

Sample size: Proposed sample size is 60 (based on Sim and Lewis, 2012 recommendations) and allowing for 20% drop-out.

Intervention: This study will use the commercially available 'Fitbit' wearable technology with its paired smartphone application. PA goals will be prescribed by a qualified, chartered physiotherapist using the American Cancer Society (ACS) guidelines (Doyle et al 2006). Participants will use the Fitbit and its paired application for 12 weeks. The Fitbit device is a tool for motivation and monitoring of PA behaviours in this intervention.

This study will also use evidence-based psychological behavioural change theory. Behavioural change techniques include 'self-monitoring of behaviour', 'goal-setting', 'feedback on behaviour' and 'information about health consequences'.

Procedures: This study includes time-points at baseline, 12 weeks (Intervention end) and 24 weeks post baseline (+/- 2 weeks (Follow-up).

Pre-intervention:Consent and PA measurement

* Consent: Study personnel meets potential participants at their outpatient appointment. The agreement of the patient's consultant to exercise has been obtained before the patient information leaflet (PIL) is provided. The researcher explains the study and gives the potential participant a consent form and a patient information leaflet and a verbal explanation of the study.
* Initial PA measurement: Participants who consent are given an Actigraph PA monitor which they will be instructed to wear for 7 days to measure their baseline physical activity levels. Participants who wish to consider the study can take the PIL home, post it back, and receive the Actigraph by post.

Baseline Session:

Participants attend

* 1) An educational session, delivered by the lead researcher, a chartered physiotherapist. This is a group information session on PA following cancer treatment.
* 2) Educational session to introduce the technological component to the participants and instruct them in use and upload of Fitbit data to allow monitoring by researcher(s).
* 3) Measurement of height, weight, BMI and body composition and 6 minute walk test During intervention. (week 1-12)
* Participants wear Fitbit and upload data for self-monitoring and monitoring by chartered physiotherapist researcher.
* Participants receive scheduled structured telephone calls, giving them feedback on their achievement of goals and reminders about uploading data as follows; 2 calls each week till week 4, 1 call a week between week 4 and 8 and 2 calls, 2 weeks apart between week 8 and week 12.

After intervention ends (12 weeks):

* Measurement of height, weight, BMI and body composition and 6 minute walk test
* Participants wear Actigraph x 7 days

  12 weeks after end of intervention:
* Measurement of height, weight, BMI and body composition and 6 minute walk test
* Participants wear Actigraph x 7 days

ELIGIBILITY:
Inclusion Criteria:

* Agreement of the participant's cancer clinician that he/she can participate, including medical clearance to exercise
* Aged >18 years
* Completed chemotherapy or radiotherapy with curative intent within the preceding 3 years. Patients may have had chemotherapy or radiotherapy as the sole treatment for cancer, but not surgery alone. Patients who are still on adjuvant hormone therapy and/or adjuvant Her2-directed therapy are eligible (with physician agreement as above).
* Able to understand English
* Owns or has access to a device which is compatible with the Fitbit app i.e. smartphone, tablet or computer.

Exclusion Criteria:

* Diagnosis of prostate cancer or upper gastro-intestinal cancer.
* Chronic medical and orthopaedic conditions that would preclude exercise (e.g uncontrolled congestive heart failure or angina, recent MI within 6 months recent Pulmonary embolism within 3 months, breathing difficulties requiring oxygen use or hospitalization, osteoarthritis causing significant mobility issues).
* Confirmed pregnancy
* Dementia, cognitive impairment or psychiatric illness that would preclude ability to participate in study.
* Incomplete haematological recovery after chemotherapy (WCC < 3, Hb < 10 or Platelets < 100).
* Patients<18 years
* Evidence of active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity (Objective) | Baseline, 12 weeks, 24 weeks
  Accelerometry will be used to monitor 7 days of activity at Week 0, Week 12 (+/- 2 weeks) and 24 weeks (+/- 2 weeks) post baseline.
Evaluation of recruitment capability and resulting sample characteristics | 12 weeks
  The number of participants we can recruit will be assessed. This will explore the potential sample size of the randomised control trial.
Data collection procedures and outcome measures | 12 weeks
  Procedures to collect data will be assessed for suitability and outcome measures used will be analysed for optimisation of measurement of clinical outcomes
Acceptability and suitability of the intervention and study procedures | 12 weeks
  Compliance with daily logging of exercise information and adherence to the intervention duration will be assessed
Use of resources and ability to manage and implement the study and intervention | 12 weeks
  The ability of study personnel and the availability of resources to implement the study will be assessed, demonstrated by successful implementation of the intervention
Preliminary evaluation of participant responses to intervention | 12 weeks
  The qualitative outcome in this feasibility study will invite participants' to provide feedback on the intervention's likelihood of being successful. Satisfaction with the technological intervention will be measured using a questionnaire given to participants at study end (12 weeks).
Change in body composition | Baseline, 12 weeks and 24 weeks
  This will be measured at baseline, 12 weeks (Intervention end) and 24 weeks post -baseline (Follow-up). This will be measured in percentage body fat.
Change in self-report PA | Baseline, 12 weeks and 24 weeks
  A modified version of the Godin Leisure Time Exercise Questionnaire will be used.
Change in quality of life | Baseline, 12 weeks and 24 weeks
  The FACT-G scale (general) (Cella et al 1993) will be used to assess quality of life.
Change in aerobic capacity/endurance | Baseline,12 weeks and 24 weeks
  This will be measured using the 6MWT (Six minute walk test).
Change in BMI | Baseline, 12 weeks and 24 weeks
  This will be measured at baseline, 12 weeks (Intervention end) and 24 weeks post -baseline (Follow-up). This will be measured in kg/m^2.
Change in Body Weight (kg) | Baseline,12 weeks and 24 weeks
  This will be measured at baseline, 12 weeks (Intervention end) and 24 weeks post -baseline (Follow-up). This will be measured in kg.
Change in waist circumference | Baseline,12 weeks and 24 weeks
  This will be measured at baseline, 12 weeks (Intervention end) and 24 weeks post -baseline (Follow-up). This will be measured in cm.
Change in quality of life | Baseline,12 weeks and 24 weeks
  The physical functional measure of the SF-36 (Brazier et al 1992) will be used to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Haberlin, BSc(Physiotherapy), Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St. James's Hospital Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Doyle C, Kushi LH, Byers T, Courneya KS, Demark-Wahnefried W, Grant B, McTiernan A, Rock CL, Thompson C, Gansler T, Andrews KS; 2006 Nutrition, Physical Activity and Cancer Survivorship Advisory Committee; American Cancer Society. Nutrition and physical activity during and after cancer treatment: an American Cancer Society guide for informed choices. CA Cancer J Clin. 2006 Nov-Dec;56(6):323-53. doi: 10.3322/canjclin.56.6.323. PMID 17135691
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Bandura, A. (1986). Social foundations of thought and action: A social cognitive theory. Englewood Cliffs, NJ, US, Prentice-Hall, Inc.
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] BALKE B. A SIMPLE FIELD TEST FOR THE ASSESSMENT OF PHYSICAL FITNESS. REP 63-6. Rep Civ Aeromed Res Inst US. 1963 Apr:1-8. No abstract available. PMID 14131272
- [Derived] Haberlin C, Broderick J, Guinan EM, Darker C, Hussey J, O'Donnell DM. eHealth-based intervention to increase physical activity levels in people with cancer: protocol of a feasibility trial in an Irish acute hospital setting. BMJ Open. 2019 Mar 8;9(3):e024999. doi: 10.1136/bmjopen-2018-024999. PMID 30852540